CLINICAL TRIAL: NCT00116610
Title: A Phase II Study of Picoplatin as Second-Line Therapy for Subjects With Resistant or Refractory Small Cell Lung Cancer
Brief Title: Picoplatin as Second-Line Therapy for Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poniard Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0402; IND No. 69,507
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-02

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; resistant; refractory; platinum; chemotherapy; second-line; relapse; sensitive
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence; Hypersensitivity | interventions — amminedichloro(2-methylpyridine)platinum(II)

INTERVENTIONS:
Drug: picoplatin

SUMMARY:
This is a Phase II research study that is designed for patients who have small cell lung cancer (SCLC) that is no longer responding to treatment. Patients will receive picoplatin, a new platinum-based agent that is currently under investigation, in 21-day cycles.

DETAILED DESCRIPTION:
Platinum drugs work by binding to DNA and preventing the rapid cell division of tumors. However, many tumors demonstrate a resistance to platinum drugs. Results from preclinical studies indicate that picoplatin (previously called AMD473 or ZD0473) may be able to overcome or partially overcome platinum resistance. More than 500 patients have received picoplatin in previous Phase I or Phase II clinical trials.

ELIGIBILITY:
Main inclusion criteria:

1. Diagnosis of small cell lung cancer.
2. Patients must have had one prior chemotherapy regimen which must have included either cisplatin or carboplatin.

[Additional eligibility criteria apply.]

Exclusion Criteria:

* Prior radiotherapy that included > 30% of the bone marrow (i.e., the whole of the pelvis or half of the spine).
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom.
* Significant heart disease.
* Uncontrolled, untreated, unstable, or symptomatic brain tumors or central nervous system disease.
* Grade 2+ peripheral neuropathy (a condition caused by damage to the nerves in the peripheral nervous system).

[Additional exclusion criteria apply.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety (outcomes will be measured approximately 1 year after the last subject has been treated)

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Breitz, MD, Study Director — Poniard Pharmaceuticals; Paul Weiden, MD, Study Director — Poniard Pharmaceuticals; David Karlin, MD, Study Director — Poniard Pharmaceuticals
Locations (55):
- United States (28):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Study Site, Los Angeles, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Eastern Connecticut Hematology/Oncology, Norwich, Connecticut
  - Oncology Hematology Group of South Florida, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - Central Georgia Hematology Oncology Associates, Macon, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Rush Medical College, Chicago, Illinois
  - Medical Center of Vincennes, Vincennes, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - The Ochsner Clinic, New Orleans, Louisiana
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - University of Missouri / Ellis Fischel Cancer Center, Columbia, Missouri
  - The Center for Cancer Care & Research, St Louis, Missouri
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - V.A. Sierra Nevada Health Care, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center Hematology/Oncology, Lebanon, New Hampshire
  - Mt. Sinai Medical Center, New York, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Consultants in Medical Oncology & Hematology, Drexel Hill, Pennsylvania
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
- Russia (25):
  - Ufa, Bashkortostan Republic
  - Stepanovskoye, Krasnogorskiy District, Moscow Oblast
  - Petrozavodsk, Republic of Karelia
  - Engel's, Saratov Oblast
  - Kazan', Tatarstan Republic
  - Izhevsk, Udmurtiya Republic
  - Cherepovets, Vologda Oblast
  - Astrakhan
  - Barnaul
  - Chelyabinsk
  - Kaliningrad
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Orenburg
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Stavropol
  - Ulyanovsk
  - Voronezh
  - Yaroslavl
  - Yekaterinburg

REFERENCES:
- [Background] Beale P, Judson I, O'Donnell A, Trigo J, Rees C, Raynaud F, Turner A, Simmons L, Etterley L. A Phase I clinical and pharmacological study of cis-diamminedichloro(2-methylpyridine) platinum II (AMD473). Br J Cancer. 2003 Apr 7;88(7):1128-34. doi: 10.1038/sj.bjc.6600854. PMID 12671715
- [Background] Douillard JY, Schiller J. ZD0473 combined with other chemotherapeutic agents for the treatment of solid malignancies. Eur J Cancer. 2002 Dec;38 Suppl 8:S25-31. doi: 10.1016/s0959-8049(02)80020-x. PMID 12645909
- [Background] Gelmon KA, Stewart D, Chi KN, Chia S, Cripps C, Huan S, Janke S, Ayers D, Fry D, Shabbits JA, Walsh W, McIntosh L, Seymour LK. A phase I study of AMD473 and docetaxel given once every 3 weeks in patients with advanced refractory cancer: a National Cancer Institute of Canada-Clinical Trials Group trial, IND 131. Ann Oncol. 2004 Jul;15(7):1115-22. doi: 10.1093/annonc/mdh278. PMID 15205207
- [Background] Gelmon KA, Vandenberg TA, Panasci L, Norris B, Crump M, Douglas L, Walsh W, Matthews SJ, Seymour LK. A phase II study of ZD0473 given as a short infusion every 3 weeks to patients with advanced or metastatic breast cancer: a National Cancer Institute of Canada Clinical Trials Group trial, IND 129. Ann Oncol. 2003 Apr;14(4):543-8. doi: 10.1093/annonc/mdg171. PMID 12649098
- [Background] Giaccone G, O'Brien ME, Byrne MJ, Bard M, Kaukel E, Smit B. Phase II trial of ZD0473 as second-line therapy in mesothelioma. Eur J Cancer. 2002 Dec;38 Suppl 8:S19-24. doi: 10.1016/s0959-8049(02)80018-1. PMID 12647701
- [Background] Gore ME, Atkinson RJ, Thomas H, Cure H, Rischin D, Beale P, Bougnoux P, Dirix L, Smit WM. Results of ZD0473 in platinum-pretreated ovarian cancer: analysis according to platinum free interval. Eur J Cancer. 2002 Dec;38 Suppl 8:S7-12. doi: 10.1016/s0959-8049(02)80014-4. PMID 12645907
- [Background] Kawamura-Akiyama Y, Kusaba H, Kanzawa F, Tamura T, Saijo N, Nishio K. Non-cross resistance of ZD0473 in acquired cisplatin-resistant lung cancer cell lines. Lung Cancer. 2002 Oct;38(1):43-50. doi: 10.1016/s0169-5002(02)00175-7. PMID 12367792
- [Background] Kanzawa F, Akiyama Y, Saijo N, Nishio K. In vitro effects of combinations of cis-amminedichloro (2-methylpyridine) platinum (II) (ZD0473) with other novel anticancer drugs on the growth of SBC-3, a human small cell lung cancer cell line. Lung Cancer. 2003 Jun;40(3):325-32. doi: 10.1016/s0169-5002(03)00072-2. PMID 12781432
- [Background] Medina-Gundrum L, Cerna C, Gomez LR, Yochmowitz M, Weitman S. AMD473 (ZD0473) exhibits marked in vitro anticancer activity in human tumor specimens taken directly from patients. Anticancer Drugs. 2003 Apr;14(4):275-80. doi: 10.1097/00001813-200304000-00004. PMID 12679731
- [Background] Murakami H, Tamura T, Yamada Y, Yamamoto N, Ueda Y, Shimoyama T, Saijo N. ZD0473 pharmacokinetics in Japanese patients: a Phase I dose-escalation study. Eur J Cancer. 2002 Dec;38 Suppl 8:S1-5. doi: 10.1016/s0959-8049(02)80012-0. PMID 12645906
- [Background] Raaphorst GP, Yang DP, Li LF, Malone S. Comparison of human tumour cell responses to cisplatin and ZD0473 with and without irradiation. Anticancer Res. 2004 Mar-Apr;24(2B):613-8. PMID 15161002
- [Background] Sharp SY, O'Neill CF, Rogers P, Boxall FE, Kelland LR. Retention of activity by the new generation platinum agent AMD0473 in four human tumour cell lines possessing acquired resistance to oxaliplatin. Eur J Cancer. 2002 Nov;38(17):2309-15. doi: 10.1016/s0959-8049(02)00244-7. PMID 12441268
- [Background] Twelves C, Reck M, Anthoney A, Gatzemeier U, Kaye S. A phase I study of ZD0473 combined with paclitaxel for the treatment of solid malignancies. Cancer Chemother Pharmacol. 2003 Oct;52(4):277-81. doi: 10.1007/s00280-003-0633-9. Epub 2003 Jun 25. PMID 12827291
- [Background] Plasencia C, Abad A, Martinez-Balibrea E, Taron M. Antiproliferative effects of ZD0473 (AMD473) in combination with 5-fluorouracil or SN38 in human colorectal cancer cell lines. Invest New Drugs. 2004 Nov;22(4):399-409. doi: 10.1023/B:DRUG.0000036682.99818.71. PMID 15292710
- [Background] Treat J, Schiller J, Quoix E, Mauer A, Edelman M, Modiano M, Bonomi P, Ramlau R, Lemarie E. ZD0473 treatment in lung cancer: an overview of the clinical trial results. Eur J Cancer. 2002 Dec;38 Suppl 8:S13-8. doi: 10.1016/s0959-8049(02)80016-8. PMID 12645908
- [Background] Gore ME, Atkinson RJ, Thomas H, Cure H, Rischin D, Beale P, Bougnoux P, Dirix L, Smit WM. A phase II trial of ZD0473 in platinum-pretreated ovarian cancer. Eur J Cancer. 2002 Dec;38(18):2416-20. doi: 10.1016/s0959-8049(02)00632-9. PMID 12460786
- See also: Poniard Pharmaceuticals website — http://www.poniard.com
- See also: CenterWatch clinical trials listings — http://www.centerwatch.com/